CLINICAL TRIAL: NCT02650817
Title: A Phase IB Study to Evaluate the Effect of RAD1901 on the Availability of Estrogen Receptor Binding Sites in Metastatic Breast Cancer Lesions Using 16α-18F-Fluoro-17β-Estradiol Positron Emission Tomography Imaging
Brief Title: Phase IB Study to Evaluate RAD1901 on the Availability of Estrogen Receptor Binding Sites in Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stemline Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAD1901-106; 2015-003555-22 (EudraCT Number); L54809.042.15 (Other: ABR nr)
Record Dates: First submitted 2016-01-06; First posted 2016-01-08 (Estimated); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — RAD1901; elacestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Elacestrant (formerly RAD1901) (Experimental): To receive daily oral elacestrant
  Interventions: Drug: RAD1901

INTERVENTIONS:
Drug: RAD1901 — RAD1901, a novel selective ER degrader (SERD)
  Other Names: Elacestrant

SUMMARY:
The purpose of this study is to visualize and quantify ER-binding sites during treatment with Elacestrant (RAD1901)

DETAILED DESCRIPTION:
The purpose of this study is to visualize and quantify ER-binding sites during treatment with Elacestrant (RAD1901) using 16α-18F-Fluoro-17β-estradiol (FES) positron emission tomography (PET) imaging

ELIGIBILITY:
Key Inclusion Criteria:

1. Patients with histologically-proven, ER-positive, human epidermal growth factor receptor 2 (HER2)-negative, locally advanced, inoperative, and/or mBC
2. Tumor progression after ≥ 6 months of at least 1 line of hormonal systemic treatment (SERM, SERD, or aromatase inhibitor) in the metastatic setting
3. Measurable disease according to Response Evaluation Criteria in Solid Tumours (RECIST) criteria v1.1 or clinically evaluable disease
4. Greater than or equal to 18 years of age
5. Patients must be post-menopausal
6. Life expectancy >3 months

Key Exclusion Criteria:

1. Greater than 3 lines of endocrine therapy for metastatic disease.
2. Prior anti-cancer treatment or investigational drug therapy within the following windows:

   1. Tamoxifen or fulvestrant therapy < 42 days before 1st 18FES-PET scan
   2. Any other anti-cancer endocrine therapy < 14 days before 1st dose of study drug
   3. Any chemotherapy < 28 days before 1st dose of study drug
   4. Any investigational drug therapy < 28 days or 3 half-lives (whichever is longer) prior to the 1st dose of study drug 2. Patients with untreated or symptomatic central nervous system (brain) metastases 3. Patients with known endometrial disorders, including evidence of endometrial hyperplasia, dysfunctional uterine bleeding, or cysts

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
Effect of ER Binding after RAD1901 treatment | 14 Days after the first dose
  To determine the effect of RAD1901 treatment on the estrogen receptor (ER) expression and estradiol binding to the ER in lesions from patients with metastatic breast cancer (mBC)

SECONDARY OUTCOMES:
Correlation of FES uptake after RAD1901 treatment to clinical response | Every 8 weeks for to up 12 months of treatment
  To determine if any changes in ER binding, as observed through FES uptake, correlate with clinical response
Tumor response will be evaluated in patients with measurable or evaluable disease, using RECISTv1.1 guidelines | Every 8 weeks for to up 12 months of treatment
  To determine if there is a tumor response to RAD1901 treatment
Safety and Tolerability assessed in terms of adverse events, serious adverse events, ECG, physical examination, ECOG performance status, vital signs, and laboratory values | Up to 30 days after the end of treatment
  Characterization of the safety of RAD1901 in this patient population
Plasma concentrations of RAD1901 will be assessed at predefined intervals | Every 28 days for up to 3 cycles
  Pharmacokinetic data will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth GE de Vries, MD, Principal Investigator — Universitair Medisch Centrum Groningen (UMCG)
Locations (5):
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - UZ Leuven Campus Gasthuisberg, Leuven
- Netherlands (3):
  - Vrije Universiteit Medisch Centrum (VUMC), Amsterdam
  - Universitair Medisch Centrum Groningen (UMCG), Groningen
  - Erasmus Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jager A, de Vries EGE, der Houven van Oordt CWM, Neven P, Venema CM, Glaudemans AWJM, Wang Y, Bagley RG, Conlan MG, Aftimos P. A phase 1b study evaluating the effect of elacestrant treatment on estrogen receptor availability and estradiol binding to the estrogen receptor in metastatic breast cancer lesions using 18F-FES PET/CT imaging. Breast Cancer Res. 2020 Sep 11;22(1):97. doi: 10.1186/s13058-020-01333-3. PMID 32912274